CLINICAL TRIAL: NCT06948383
Title: Serratus Posterior Superior Intercostal Plane Block Versus Serratus Anterior Plane Block for Breast Surgery: A Randomized Controlled Trial
Brief Title: SPSIPB vs. SAPB in Breast Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Merve Sena BAYTAR, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/01-12
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain; Quality of Recovery
Keywords: postoperative pain; pain scores; Pain management; Fasial plane blocks
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (No Intervention)
- Group SPSIPB (Active Comparator)
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block
- Group SAPB (Active Comparator)
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block — administer 30 mL %0.25 bupivacain between third costa and serratus posterior superior muscle
  Arms: Group SPSIPB
Procedure: Serratus Anterior Plane Block — administer 30 mL %0.25 bupivacain between 5th costa and serratus anterior muscle in midaxiller line
  Arms: Group SAPB

SUMMARY:
The effects of the newly defined serratus posterior superior intercostal plane block and serratus anterior plane block on postoperative analgesia and quality of recovery in women undergoing breast surgery will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received informed consent form Patients who will undergo Breast Cancer Surgery aged between 18-65

Exclusion Criteria:

* <18 years and >65 years
* ASA ≥ IV
* History of allergy to local anesthetics
* Clinical diagnosis of coagulation disorders
* Infection near the entry site
* Chronic analgesic use Patients who will undergo bilateral Breast Cancer Surgery
* Body mass index >35
* Clinical diagnosis of Dementia or confusion
* Lack of cooperation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | up to 24 hour after surgery
  total opioid consumption during postoperative 24 hours

SECONDARY OUTCOMES:
Postoperative pain scores | postoperative 2nd 6th, 12th 24th hour
  Pain scores evaluate with Numeric rating scale. 0= no pain, 10= unbearable pain
quality of recovery | postoperative 24 hour
  Recovery quality will be measured with Quality of recovery-15 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No